CLINICAL TRIAL: NCT04190043
Title: Womens's Experiences of Pregnancy Loss Aftercare in the Gynecological Emergency Department of Montpellier Hospital.
Brief Title: Womens's Experiences of Pregnancy Loss Aftercare in the Gynecological Emergency
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0547
Record Dates: First submitted 2019-12-04; First posted 2019-12-09 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Miscarriage
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction: Scientific papers on the womens's experiences of pregnancy loss aftercare in the emergency department show that how announcement is made and how much caregivers show empathy to women, help women to face this difficult moment. However, in most studies, women say they did not have enough information nor support from the medical teams.

Diagnosis of miscarriage in the emergency department is the routine for the caregiver but is often experienced by the woman as the loss of a child.

This study has for goal to bring to light the discrepancy between the caregivers's experience and the women's experience :the given information, the time for consultation, the empathy.

Methods : 2 months after the diagnosis of miscarriage in the emergency room, patients receive a phone call with explanations about the project. If the patient gives her consent, she receives a computer questionnaire by email (questions about : reasons for coming to the emergency room, circumstances of announcement, information given in the emergency room, satisfaction with the care…) In parallel, caregivers have to complete a questionnaire about the same parameters.

The main objective of this study is to evaluate womens's experiences of pregnancy loss aftercare in the emergency department of Montpellier Hospital.

The second objective is to assess the discrepancy between the patient's experience and the caregivers' experience in this situation with the aim of suggesting improvement.

ELIGIBILITY:
Inclusion criteria :

An individual must fulfill all of the following criteria in order to be eligible for study enrollment:

* Women > 18 years old
* French speaker
* Diagnosis and management of miscarriage / pregnancy loss in the emergency department
* Miscarriage / pregnancy loss < 15 SA

Exclusion criteria:

* Subject unable to read or/and write
* Pregnancy loss > 15 SA.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with diagnosis of pregnancy loss in the gynecological emergency department of Montpellier Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
to evaluate womens's experiences of pregnancy loss aftercare | 1 day
  Computer questionnaire (Patient characteristics, Reason for coming to the emergency room, Circumstances of the announcement, Information given to the emergency room, Reception in emergencies) with Patient satisfied or not with the care in emergencies department: 0 -> 5

SECONDARY OUTCOMES:
evaluate the discrepancy between the patient's experience and the caregivers' experience in front of diagnosis of miscarriage. | 1 day
  Computer questionnaire for the caregivers (Circumstances of the announcement, Information given to the emergency room, Reception in emergencies)

CONTACTS AND LOCATIONS:
Overall Officials: Clara Compan, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC